CLINICAL TRIAL: NCT00880074
Title: Early Prediction of Clinical Response to Chemotherapy With FLT-PET
Brief Title: FLT-PET in Predicting Response to Chemotherapy in Patients With Advanced Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2008-0106; NCI-2012-01625 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCI-2010-01046; 2008-0106 (Other: M D Anderson Cancer Center); NCI-2012-01625 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2009-04-09; First posted 2009-04-13 (Estimated); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Malignant Neoplasm
MeSH Terms: conditions — Neoplasms | interventions — alovudine; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Diagnostic (fluorine F-18 fluorothymidine PET) (Experimental): Patients undergo fluorine F-18 fluorothymidine PET at baseline, at day 6-8 of course 1, day 20 of course 2, and prior to day 1 of course 3.
  Interventions: Drug: Fluorothymidine F-18; Other: Laboratory Biomarker Analysis; Procedure: Positron Emission Tomography

INTERVENTIONS:
Drug: Fluorothymidine F-18 — Undergo fluorine F-18 fluorothymidine PET
  Other Names: 18F-FLT; 3'-Deoxy-3'-(18F) Fluorothymidine; 3'-deoxy-3'-[18F]fluorothymidine; ALOVUDINE F-18; Fluorothymidine F 18
Other: Laboratory Biomarker Analysis — Optional correlative studies
Procedure: Positron Emission Tomography — Undergo fluorine F-18 fluorothymidine PET
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT

SUMMARY:
This clinical trial studies fluorine F-18 fluorothymidine (FLT)-positron emission tomography (PET) in predicting response to chemotherapy in patients with advanced malignancies. FLT solution can help locate cancer cells inside the body. Diagnostic procedures, such as FLT-PET, may help find tumors and measure a patient's response to treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if concurrent treatment with temsirolimus and bevacizumab demonstrates a dose-dependent decrease in FLT-PET standardized uptake value which correlates with clinical response.

SECONDARY OBJECTIVES:

I. To determine the relationship between FLT-PET and markers of angiogenesis and drug activity in tumor biopsy, along with surrogate peripheral blood markers of target inhibition and drug activity.

OUTLINE:

Patients undergo fluorine F-18 fluorothymidine PET at baseline, at day 6-8 of course 1, day 20 of course 2, and prior to day 1 of course 3.

ELIGIBILITY:
Inclusion Criteria:

* Patients actively enrolled and being treated on protocol 2007-0668: Combination Therapy with Bevacizumab and Temsirolimus in Patients with Advanced Malignancy at M.D. Anderson Cancer Center; these patients must have met the inclusion and exclusion criteria for that protocol
* Women of child-bearing potential (as defined as women who are not post-menopausal for 12 months or who have had no previous surgical sterilization) and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 90 days after the last dose
* Ability to understand and the willingness to sign a written informed consent document
* Patient actively enrolled and being treated on protocol 2012-0061 "A Phase I Trial of Bevacizumab, Temsirolimus Alone and in Combination with Valproic Acid or Cetuximab in Patients with Advanced Malignancy" at M.D. Anderson Cancer Center

Exclusion Criteria:

* Pregnant or breast-feeding women
* History of hypersensitivity to 3'-deoxy-3'-18F-fluorothymidine (18F-FLT) or any component of the formulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-04-09 (Actual); Primary Completion 2022-02-04 (Actual); Study Completion 2022-02-04 (Actual)

PRIMARY OUTCOMES:
Response to Chemotherapy Shown in FLT-PET Scans | through study completion; an average of 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Sarina A Piha-Paul, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org